CLINICAL TRIAL: NCT03057249
Title: The Impact of a Selected Surgical Procedure on Skin Blood Perfusion of the Abdominal Wall Evaluated by Dynamic Infrared Thermography (DIRT)
Brief Title: Skin Perfusion After Abdominal Surgery
Acronym: DIRTSURGERY
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/176
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2017-02

CONDITIONS: Surgical Wound Infection
Keywords: Surgery; Thermography; Perfusion; Imaging
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dynamic infrared thermography (DIRT) — Evaluating abdominal skin perfusion with DIRT

SUMMARY:
The purpose of this study is to evaluate the consequences of 3 selected surgical procedures on abdominal wall perfusion in order to help to reduce postoperative complication related to inadequate tissue perfusion. The selected surgical procedures are a) abdominoplasty, b) breast reconstruction with a free flap from the lower abdomen and c) endovascular stenting of an abdominal aorta aneurism. These operations are all standard surgical procedures frequently performed at the University Hospital of North Norway, Tromsø. The abdominal wall perfusion will be evaluated with the use of Dynamic Infrared Thermography (DIRT).

DETAILED DESCRIPTION:
Introduction Wound healing problems after surgery are a stressful experience for patients. Wound dressing changes are often on a daily basis and can cause considerable discomfort to the patient as these are often painful. Wound healing problems can lead to complications like wound infection, hernia formation, wound rupture or even tissue necrosis. These complications are often associated with prolonged hospital stays and reoperations and cause an economic burden to the hospital health budget. It is generally accepted that adequate blood perfusion of the wound edges is required for optimal wound healing. Greater understanding of the impact of a surgical procedure on skin perfusion may help to reduce postoperative wound healing problems. Such will have great clinical relevance.

Aim Can postoperative wound complications involving the abdominal wall be explained by changes in skin blood perfusion?

Main results from the literature study In surgery, knowledge on the vascular anatomy is applied in order to place incisions in such a manner that a good approach is combined with minimal damage to the vascular anatomy. Knowledge on vascular anatomy does not provide exact information on how skin perfusion alters after surgery. The invasive method indocyanine green fluorescence-agiography (ICG-FA) can be used to evaluate intraoperatively the effect of an abdominoplasty on skin perfusion. However, animal studies in flap surgery have clearly shown that tissue perfusion is a dynamic process. Using dynamic infrared thermography (DIRT) in a clinical setting revealed that flap perfusion is a dynamic process that takes place over days during the postoperative phase. DIRT is a non-invasive technique that relies on measuring skin surface temperatures. Studies have shown that there is a close correlation between skin temperature and skin perfusion. DIRT has been shown to be a good alternative to ICF-FA to visualize skin perfusion.

Purpose of the study The purpose of the study is to analyze the impact of a surgical procedure on skin perfusion of the abdominal wall in order to increase our understanding on how postoperative wound healing problems can be avoided.

Study population The study population will include patients that are undergoing one of the following operations; a) abdominoplasty, b) breast reconstruction after breast cancer with a free flap from the lower abdomen and c) endovascular stenting of the abdominal aorta for aneurysm. These surgical procedures are frequently performed procedures at the University Hospital of North Norway (UNN). Based on the vascular anatomy of the abdominal wall, each procedure will have an impact on the skin perfusion of the abdominal wall.

Material and Methods Approval will be obtained from the regional ethical committee and the principles outlined in the Declaration of Helsinki will be followed.

Study I The inclusion criteria are patients scheduled for abdominoplasty who are non-smokers or have stopped smoking at least 3 months prior to surgery and have no supraumbilical abdominal scars from previous surgery Study II The inclusion criteria are patients scheduled for secondary unilateral free abdominal flap breast reconstructions who are non-smokers or have stopped smoking at least 3 months prior to surgery and have no abdominal scar from previous surgery.

Study III Patients who are scheduled for endovascular stenting of the abdominal aorta.

DIRT will be performed on the day before surgery, intraoperatively and on the 1st, 3rd and 6th postoperative day with all DIRT examinations performed in the same supine position for study I and II. For study III, the same protocol will be used, however, no intraoperative DIRT examination will be performed. For study III, thermal images are taken from both lower extremities during the abdominal DIRT examination to see if stenting causes a change in rewarming of the lower extremities following stenting.

An IR camera (FLIR ThermaCAM S65 HS FLIR Systems, FLIR Systems AB, Boston, MA) will be positioned directly above the exposed anterior thorax and abdomen. This camera can produce sequences of high-definition digital IR images with an accuracy of 0.1º C. Thermal emissivity is set to 0.98 and the accuracy of the camera will be regularly checked against a black body with a traceable temperature source (Model IR-2103/301, Infrared Systems Development Corp., Florida, USA). IR images are taken at regular intervals to register the rate and pattern of skin recovery for 3 minutes after a mild cold challenge. Images are electronically stored and afterwards processed using image analysis software ThermaCAM Researcher Pro 2.8 SR-1 (FLIR Systems AB).

The pre- and postoperative images are taken in a dedicated laboratory (room temperature 21-23°C) before and during recovery following a cold challenge after an acclimatization period of 10 minutes with the thoracic and abdominal wall exposed. The thermal challenge is delivered by blowing air at room temperature over the skin surface for 2 minutes with a desktop fan. The intraoperative examination is performed with the patient in general anaesthesia just before and at the end of surgery. The thermal cold challenge is performed by washing the thorax and abdomen evenly for 1 minute with gauze soaked in saline at room temperature (22-23°C).

The abdomen is divided into vascular zones as defined by Huger. The mean skin temperature is calculated for each zone in the postoperative phase before cooling, at end cooling and at 1, 2 and 3 minutes recovery. A qualitative analysis of the changes of pattern and rate of recovery of hot spots within each zone is made and compared with the results from the other zones. A one tailed t test for paired variables is use to see if there is a statistically significant in the mean temperatures between zones at each time point of rewarming. Statistical significance is defined as p<0.05.

Publications The results from each study will be published in an international peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for

1. Abdominoplasty
2. DIEP breast reconstruction
3. Aorta stenting

Exclusion Criteria:

Surgery not indicated Smokers

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for
  1. Abdominoplasty
  2. DIEP breast reconstruction
  3. Aorta stenting
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Perfusion dynamics following surgical procedures | First five postoperative days
  DIRT findings on the abdominal wall after three different types of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Louis de Weerd, MD PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No
The study is based on qualitative evaluation of individual thermographic images that are not suitable for public sharing

REFERENCES:
- [Result] Nahai F, Brown RG, Vasconez LO. Blood supply to the abdominal wall as related to planning abdominal incisions. Am Surg. 1976 Sep;42(9):691-5. No abstract available. PMID 133628
- [Result] Boltz MM, Hollenbeak CS, Julian KG, Ortenzi G, Dillon PW. Hospital costs associated with surgical site infections in general and vascular surgery patients. Surgery. 2011 Nov;150(5):934-42. doi: 10.1016/j.surg.2011.04.006. Epub 2011 Jun 15. PMID 21676424
- [Result] Broex EC, van Asselt AD, Bruggeman CA, van Tiel FH. Surgical site infections: how high are the costs? J Hosp Infect. 2009 Jul;72(3):193-201. doi: 10.1016/j.jhin.2009.03.020. Epub 2009 May 31. PMID 19482375
- [Result] Hunt TK, Hopf H, Hussain Z. Physiology of wound healing. Adv Skin Wound Care. 2000 May-Jun;13(2 Suppl):6-11. PMID 11074996
- [Result] Sen CK. Wound healing essentials: let there be oxygen. Wound Repair Regen. 2009 Jan-Feb;17(1):1-18. doi: 10.1111/j.1524-475X.2008.00436.x. PMID 19152646
- [Result] Huger WE Jr. The anatomic rationale for abdominal lipectomy. Am Surg. 1979 Sep;45(9):612-7. PMID 159651
- [Result] Mayr M, Holm C, Hofter E, Becker A, Pfeiffer U, Muhlbauer W. Effects of aesthetic abdominoplasty on abdominal wall perfusion: a quantitative evaluation. Plast Reconstr Surg. 2004 Nov;114(6):1586-94. doi: 10.1097/01.prs.0000138757.33998.ee. PMID 15509954
- [Result] Dhar SC, Taylor GI. The delay phenomenon: the story unfolds. Plast Reconstr Surg. 1999 Dec;104(7):2079-91. doi: 10.1097/00006534-199912000-00021. PMID 11149772
- [Result] de Weerd L, Miland AO, Mercer JB. Perfusion dynamics of free DIEP and SIEA flaps during the first postoperative week monitored with dynamic infrared thermography. Ann Plast Surg. 2009 Jan;62(1):42-7. doi: 10.1097/SAP.0b013e3181776374. PMID 19131718
- [Result] de Weerd L, Mercer JB, Weum S. Dynamic infrared thermography. Clin Plast Surg. 2011 Apr;38(2):277-92. doi: 10.1016/j.cps.2011.03.013. PMID 21620152